CLINICAL TRIAL: NCT04359498
Title: Retrospective Study of Surgical Complications in Patients With Defunctioning Stoma After Low Anterior Resection for Rectal Cancer
Brief Title: Retrospective Study of Surgical Complications in Patients With Defunctioning Stoma After Low Anterior Resection (LAR)
Status: Completed | Type: Observational
Sponsor: Safeheal (Industry)
Collaborators: Clinical Research Consultants, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SH-001
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Rectal Cancer
Keywords: Low Anterior Resection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LAR for rectal cancer: Retrospective chart review for surgical complications related to the LAR surgery, the stoma (diverting loop ileostomy) creation and the stoma reversal procedure after LAR for rectal cancer.

SUMMARY:
This study is being conducted to evaluate the incidence and type of surgical complications occurring in patients who have a defunctioning stoma after LARfor rectal cancer. The data from this retrospective study will be analyzed by the study Sponsor to aid in designing a prospective clinical trial for a new technology that offers a treatment alternative to standard of care defunctioning stoma in patients undergoing LAR for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18 years of age or older at the time the LAR surgery was performed.
2. Having an open or minimally invasive colorectal resection with diverting loop ileostomy surgical procedure performed between January 15, 2015 and January 15, 2019 for treatment of a known or suspected malignant condition.
3. Availability of medical records for a postoperative visit occurring 12 months (± 3 months) after the LAR surgery.

Exclusion Criteria:

1. Planned surgical procedure is a Hartmann's procedure (surgical resection of the rectosigmoid colon with closure of the anorectal stump and formation of an end colostomy).
2. Having a documented medical history of inflammatory bowel disease prior to the LAR surgery.
3. Having a concomitant major surgical procedure performed in combination with the LAR surgery (e.g., colorectal resection with hepatectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent LAR for rectal cancer and are 12 months or longer postoperative from the LAR surgery will be reviewed for eligibility.
Sampling Method: Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Surgical complications | 12 Months
  Characterize the type and incidence of surgical complications related to the LAR, the stoma creation and the stoma reversal after LAR for rectal cancer.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - University of California, Irvine, Irvine, California
  - Keck School of Medicine of USC, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of South Florida, Tampa, Florida
  - UMASS Memorial, Worcester, Massachusetts
  - Northwell Health, Inc., New Hyde Park, New York
  - Icahn School of Medicine, New York, New York
- Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No